CLINICAL TRIAL: NCT04789135
Title: Evaluation of Response to Use of Intravesical Ozone Gas in Interstitial Cystitis/Bladder Pain Syndrome
Brief Title: Evaluation of Response to Use of Intravesical Ozone Gas in Interstitial Cystitis /Bladder Pain Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Anhembi Morumbi University (Other)
Responsible Party: Principal Investigator, Maria Verônica de Araújo Pires, Master's Student, Anhembi Morumbi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVdeAraujoPires
Record Dates: First submitted 2021-03-01; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Interstitial Cystitis, Chronic; Bladder Pain Syndrome
Keywords: Interstitial cystitis; Bladder pain Sydrome; Ozone therapy
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Ozone

STUDY DESIGN:
Intervention Model Description: Experimental. Nature of descriptive analysis of the exploratory type, as it seeks to gather characteristics and information about the studied phenomena
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ozone Therapy (Experimental): Administration of intravesical ozone gas in patients with Interstitial cystitis/bladder pain sydrome
  Interventions: Drug: Ozone

INTERVENTIONS:
Drug: Ozone — Treatment consists of direct instillation into the bladder of ozone gas, with concentration of 20µg / ml - 60ml via urethral catheter.
  Other Names: Ozone Therapy; Intravesical medications

SUMMARY:
Interstitial Cystitis / bladder pain syndrome (CI / BPS) is a debilitating pathology with a negative impact on the quality of life of affected individuals. It is characterized as the sensation of pain or discomfort related to the urinary bladder, accompanied by symptoms of the lower urinary tract, in the absence of infection. Among the phenotypes are Cystitis with Hunner's ulcer, essentially inflammatory pathology and without Hunner's lesion, non-inflammatory frequently associated with somatoform systemic changes. Functional changes in urothelium and epithelial barrier, neurogenic inflammation and autoimmune mechanisms are involved in the development of the disease.

Medical ozone has anti-inflammatory, antioxidant, cytoprotective, antimicrobial and immunomodulatory properties. When administered, it is dissolved in biological fluids, immediately reacting with glycoproteins composed of carbohydrates and polypeptide chains. This reaction results in the formation of hydrogen peroxide (H2O2), lipid oxidation products (LOS), increased activation of erythroid-related nuclear transcription factors (Nrf2) activation of antioxidant response transcription elements (ARE) and increased variety of antioxidant enzymes that act as free radical scavengers. Benefits of O3 have been demonstrated in the treatment of neuropathic pain and hyperalgesia associated with the analgesic and anti-inflammatory effect.

The objective of this work is to evaluate the effect of intravesical ozone gas administration in patients with Interstitial Cystitis / Painful Bladder Syndrome with low response to conventional therapy.

DETAILED DESCRIPTION:
Interstitial Cystitis / bladder pain syndrome (IC / BPS) is a debilitating pathology with a negative impact on the quality of life of patients. According to the European Society for the Study of IC / BPS (ESSIC) it is expressed as a sensation of pain, pressure or discomfort related to the urinary bladder accompanied by symptoms of the lower urinary tract. Symptoms occur in the absence of infection and obvious pelvic pathologies lasting more than six weeks.

The CI / BPS has a variety of clinical phenotypes and potential etiologies. Among the phenotypes are included cystitis (IC) associated with Hunner's ulcers, known as ESSIC BPS type 3 and without Hunner's lesion, ESSIC type 1,2. Differentiation between the sub-types is performed through cystoscopy by the presence or absence of Hunner's lesions.

The dysfunctions resulting from IC / BPS originate around the bladder, adjacent pelvic organs and part of the neural tissue that controls bladder function. Functional changes in urothelium and epithelial barrier, neurogenic inflammation and autoimmune mechanisms are involved in the development of the disease.

The urothelium is covered by a layer of glycosaminoglycans (GACs) forming a protective barrier to the underlying tissues against urinary constituents and promoting selective control of molecules towards the bladder wall.

Molecular and structural changes in the GACs layer associated with the inflammatory process cause changes in urothelial permeability allowing toxic substances and urinary cations to reach the muscle and neural layer. The loss of the urothelial barrier allows chemical, cytotoxic stimuli to come into direct contact with peripheral bladder afferent neurons with persistent sensitization, central nervous amplification and local inflammatory reaction.

Neurotransmitters released by peripheral neurons, including vasoactive peptides, calcitonin and tachykinins induce mast cell degranulation and release of pro - inflammatory mediators such as histamine, serotonin, tryptase, TNF-α and NGF, IL6 resulting in local inflammation. These inflammatory mediators act on afferent neurons in a positive feedback loop resulting in the release of neurotransmitters that exacerbate mast cell degranulation and local inflammatory response, with functional destruction of bladder tissue, fibrosis, low Detrusor compliance and hyperactivity.

Alterations in the Autonomic Nervous System with sympathetic hyperactivity and exacerbation of the sensation of pain induces a condition of hyperalgesia associated with stress, in addition to contributing to the maintenance and worsening of the functional changes of the bladder. Persistent spinal cord activation can mediate pain after resolution of the inflammatory process.

The bladder pain syndrome is a common cause of chronic pelvic pain. It presents low long-term therapeutic response, innovative therapeutic modalities in the field of current studies.

Ozone gas (O3) is a molecule made up of three oxygen atoms with an unstable structure given a mesomeric effect. It has an average life of 40min at 20º C.

The interest in the therapeutic use of O3 in several diseases is growing. This interest is associated with anti-inflammatory, cytoprotective, antioxidant, antimicrobial and immunomodulatory properties. Animal models suggest beneficial and prophylactic effects of O3 therapy on age-related oxidative stress.

When administered, O3 is dissolved in biological fluids, reacting immediately with glycoproteins composed of carbohydrates and polypeptide chains (proteoglycans, collagen types II and IV). This reaction results in the formation of hydrogen peroxide (H2O2), lipid oxidation products (LOS), increased activation of erythroid-related nuclear transcription factors (Nrf2) activation of antioxidant response transcription elements (ARE) and increased variety of antioxidant enzymes that act as free radical scavengers.

Benefits of O3 have been demonstrated in the treatment of neuropathic pain and hyperalgesia associated with the analgesic and anti-inflammatory effect. Animal models demonstrate decreased and normalized expression of caspases and IL -1β, TNF. At low doses, O3 reduces the synthesis of prostaglandins (PGS) by inhibiting prostaglandin endoperoxide synthase (PGHS2) and cyclooxygenase (COXs). This fact is critical in preventing neural sensitization following persistent stimulation of intracellular pathways responsible for the excessive release of cytokines, PGs, or glutamate.

ETHICAL CRITERIA. All patients must undergo the signature of the Informed Consent Form for Medical Treatment with Medicinal Ozone METHODOLOGY This is an interventional, controlled study that provides for the application of intravesical ozone gas as an alternative treatment for patients with interstitial cystitis/bladder pain syndrome The study foresees the participation of 50 patients with interstitial cystitis /bladder pain syndrome and will be developed in the Hospital Unit of Nephrology and Urology Distal, located in the city of Jacareí, São Paulo, Brazil.

DIAGNOSTIC CRITERIA 1.1 History A thorough general medical history to identify typical diagnostic symptoms of Interstitial cystitis and bladder pain syndrome and other potential mimicking causative conditions. Figure 1 shows a flowchart of clinical approach.

1.2 Physical examination The physical exam include an abdominal and pelvic exam, with particular focus for masses, bladder distension and suprapubic tenderness. In men, sensitivity will be analyzed through palpation of the perineal area between the scrotum and anus. In women sensitivity will be analyzed through palpation of the anterior vaginal wall along the course of the urethra up to the bladder neck.

1.3 DIAGNOSTIC METHODS A. Urinalysis and Culture A urine dipstick will be performed on all patients The laboratory method of qualitative and quantitative determination of pathogenic microorganisms in the urinary tract will be performed. Urinary tract infection will be characterized by the bacterial growth of at least 105 Colony Forming Units per ml of urine (100.000 CFU / mL). The collection of urinary sample will be performed with aseptic technique avoiding contamination with the microbiota of the perineum, prostate, urethra and vagina.

B. Ultrasound Urinary Tract Abdominal and pelvic ultrasonography will be performed on all patients. C. Urodynamic Assessment Study carried out with the purpose of obtaining functional information on vesical storage and emptying.

D Symptom scores Symptom score IC / BPS will be used to establish a baseline of symptom severity at admission and subsequently, track response to treatment and disease relapse. It Will be used in the O'Leary-Sant Symptom and Problem Index, that is validated and widely used as a self-report measure of urinary and pain symptoms and how problematic these symptoms are for individuals. The measure assesses both symptoms and problems of IC/BPS each with four questions, yielding a symptom score (ICSI), problem score (ICPI), and total severity score. Symptom scores (ICSI) range from 0 to 21 and problem scores (ICPI) range from 0 to 16, with a total ICSI/ICPI combined score ranging from 0 to 37[21].

TREATMENT PROTOCOL Patients who meet inclusion criteria will be subjected to conventional treatment of the diagnoses made and submitted to the application of intravesical medicinal ozone gas.

Therapeutic Scheme

1° Bladder wash with 0.9% Saline - 500 ml performed through urethral tube n° 10; 2° Bladder emptying ; 3° Medical Ozone gas infusion 20 µg / ml - 60ml, intravesical forecast of two weekly sessions, with a total of six applications.

Clinical Follow-up Patients will be evaluated at each session using the score IC/BPS and possible side effects. At the end of the sixth session, Uroculture and Urofluxometry will be scheduled.

Monthly assessments will be scheduled for up to six months from the end of treatment to verify the maintenance of therapeutic response over time DATA ANALYSIS Qualitative data will be grouped into categories followed by the corresponding percentage. The analysis will be performed using SPSS software and Microsoft Excel.

Quantitative data will be presented in frequency distribution tables with mean, median and descriptive statistics. Statistical analysis performed using Student's t-test with significance values p> 0.05.

CLINICAL RISK It is a risk procedure estimated as small since the administration of Ozone with controlled doses is safe and determinant of small side effects. The discomfort caused by the use of the urethral tube is small and performed safely.

The specialized professionals who will conduct the experiments will be available and able to offer any necessary attention BENEFIT Patients who will be included in the present study have chronic pathology with impaired quality of life and inadequate response to conventional therapy. Based on scientific evidence, Ozone Therapy is expected to be a treatment alternative.

ELIGIBILITY:
Inclusion Criteria:

* Interstitial Cystitis
* Bladder pain Syndrome

Exclusion Criteria:

* Malignant Neoplasm
* Bladder Lithiasis.
* Lower Tract Infections

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the response to the use of intravesical medicinal ozone gas in patients with Interstitial Cystitis / Bladder Pain Syndrome (IC / BPS) using the O'Leary Sant Symptom and Problem Index questionnaire | The O'Leary Sant Symptom and Problem Index questionnaire will be applied upon admission, after the third and sixth application of intravesical. Follow-up will be carried out monthly thereafter until the sixth month of the intervention as a response check
  The O 'Leary Sant Symptom and Problem Index is validated as a self-report measure of urinary symptoms and pain and how problematic these symptoms are for individuals with IC / BPS. The measure assesses symptoms and problems of IC / BPS through four questions, generating a symptom score (ICSI), problem score (ICPI) and total severity score. Symptom scores (ICSI) range from 0 to 21 and problem scores from 0 to 16, with a combined total score of 0 to 37. ICSI and ICPI score values greater than 6 alone are considered severe symptoms. Symptom scores (ICSI) greater than 5 have 94% sensitivity and 50% specificity for the diagnosis of patients with IC / BPS.
  At the end of the study, the symptom score cut-off point (ICSI) below 5 will be considered as a therapeutic response measure. The problem scores will be assessed through an improvement percentage, with values greater than 75% being considered as adequacy.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Pires, Pires, Principal Investigator — Anhembi Morumbi University
Locations (1):
- Distal Nefrologia e Urologia, Jacareí, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The study aims to publicly share the untreated data of the individuals evaluated, provided that, with due regard for the premise of preserving patient identification, assumed in the Informed Consent Form for Medical Treatment with Medicinal Ozone.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be shared within a maximum period of six months from the date of publication of the trial

REFERENCES:
- [Background] Akiyama Y, Luo Y, Hanno PM, Maeda D, Homma Y. Interstitial cystitis/bladder pain syndrome: The evolving landscape, animal models and future perspectives. Int J Urol. 2020 Jun;27(6):491-503. doi: 10.1111/iju.14229. Epub 2020 Apr 4. PMID 32246572
- [Background] Grover S, Srivastava A, Lee R, Tewari AK, Te AE. Role of inflammation in bladder function and interstitial cystitis. Ther Adv Urol. 2011 Feb;3(1):19-33. doi: 10.1177/1756287211398255. PMID 21789096
- [Background] Akiyama Y, Hanno P. Phenotyping of interstitial cystitis/bladder pain syndrome. Int J Urol. 2019 Jun;26 Suppl 1:17-19. doi: 10.1111/iju.13969. PMID 31144756
- [Background] Birder LA. Pathophysiology of interstitial cystitis. Int J Urol. 2019 Jun;26 Suppl 1:12-15. doi: 10.1111/iju.13985. PMID 31144735
- [Background] Quaghebeur J, Wyndaele JJ. Bladder pain syndrome (BPS): Symptom differences between type 3C BPS and non-type 3C BPS. Scand J Urol. 2015;49(4):319-20. doi: 10.3109/21681805.2014.982170. Epub 2014 Nov 27. No abstract available. PMID 25428753
- [Background] Han E, Nguyen L, Sirls L, Peters K. Current best practice management of interstitial cystitis/bladder pain syndrome. Ther Adv Urol. 2018 Mar 19;10(7):197-211. doi: 10.1177/1756287218761574. eCollection 2018 Jul. PMID 30034539
- [Background] Arance I, Ramon de Fata F, Angulo JC, Gonzalez-Enguita C, Errando C, Cozar JM, Esteban M. [Available evidence about efficacy of different restoring agents of glycosaminoglycans for intravesical use in interstitial cystitis]. Actas Urol Esp. 2013 Feb;37(2):92-9. doi: 10.1016/j.acuro.2012.10.002. Epub 2012 Dec 20. Spanish. PMID 23260184
- [Background] Patnaik SS, Lagana AS, Vitale SG, Buttice S, Noventa M, Gizzo S, Valenti G, Rapisarda AMC, La Rosa VL, Magno C, Triolo O, Dandolu V. Etiology, pathophysiology and biomarkers of interstitial cystitis/painful bladder syndrome. Arch Gynecol Obstet. 2017 Jun;295(6):1341-1359. doi: 10.1007/s00404-017-4364-2. Epub 2017 Apr 8. PMID 28391486
- [Background] Sagai M, Bocci V. Mechanisms of Action Involved in Ozone Therapy: Is healing induced via a mild oxidative stress? Med Gas Res. 2011 Dec 20;1:29. doi: 10.1186/2045-9912-1-29. PMID 22185664
- [Background] Smith NL, Wilson AL, Gandhi J, Vatsia S, Khan SA. Ozone therapy: an overview of pharmacodynamics, current research, and clinical utility. Med Gas Res. 2017 Oct 17;7(3):212-219. doi: 10.4103/2045-9912.215752. eCollection 2017 Jul-Sep. PMID 29152215
- [Background] Di Mauro R, Cantarella G, Bernardini R, Di Rosa M, Barbagallo I, Distefano A, Longhitano L, Vicario N, Nicolosi D, Lazzarino G, Tibullo D, Gulino ME, Spampinato M, Avola R, Li Volti G. The Biochemical and Pharmacological Properties of Ozone: The Smell of Protection in Acute and Chronic Diseases. Int J Mol Sci. 2019 Feb 1;20(3):634. doi: 10.3390/ijms20030634. PMID 30717203
- [Background] Fuccio C, Luongo C, Capodanno P, Giordano C, Scafuro MA, Siniscalco D, Lettieri B, Rossi F, Maione S, Berrino L. A single subcutaneous injection of ozone prevents allodynia and decreases the over-expression of pro-inflammatory caspases in the orbito-frontal cortex of neuropathic mice. Eur J Pharmacol. 2009 Jan 28;603(1-3):42-9. doi: 10.1016/j.ejphar.2008.11.060. Epub 2008 Dec 6. PMID 19100257
- [Background] Wei A, Feng H, Jia XM, Tang H, Liao YY, Li BR. Ozone therapy ameliorates inflammation and endometrial injury in rats with pelvic inflammatory disease. Biomed Pharmacother. 2018 Nov;107:1418-1425. doi: 10.1016/j.biopha.2018.07.137. Epub 2018 Sep 1. PMID 30257358
- [Background] Elvis AM, Ekta JS. Ozone therapy: A clinical review. J Nat Sci Biol Med. 2011 Jan;2(1):66-70. doi: 10.4103/0976-9668.82319. PMID 22470237
- [Background] Hernandez FA. To what extent does ozone therapy need a real biochemical control system? Assessment and importance of oxidative stress. Arch Med Res. 2007 Jul;38(5):571-8. doi: 10.1016/j.arcmed.2007.03.002. PMID 17560465
- [Background] Uguz S, Demirer Z, Uysal B, Alp BF, Malkoc E, Guragac A, Turker T, Ates F, Karademir K, Ozcan A, Yildirim I, Korkmaz A, Guven A. Medical ozone therapy reduces shock wave therapy-induced renal injury. Ren Fail. 2016 Jul;38(6):974-81. doi: 10.3109/0886022X.2016.1172941. Epub 2016 Apr 20. PMID 27099130
- [Background] 19. Renate Viebahn-Hänsler , Olga Sonia León Fernández & Ziad Fahmy (2012) Ozone in Medicine: The Low- Dose Ozone Concept-Guidelines and Treatment Strategies, Ozone: Science & Engineering: The Journal of the International Ozone Association, 34:6, 408-424, DOI: 10.1080/01919512.2012.717847
- [Background] McKernan LC, Bonnet KR, Finn MTM, Williams DA, Bruehl S, Reynolds WS, Clauw D, Dmochowski RR, Schlundt DG, Crofford LJ. Qualitative Analysis of Treatment Needs in Interstitial Cystitis/Bladder Pain Syndrome: Implications for Intervention. Can J Pain. 2020;4(1):181-198. doi: 10.1080/24740527.2020.1785854. Epub 2020 Sep 1. PMID 33367196
- [Result] Malde S, Palmisani S, Al-Kaisy A, Sahai A. Guideline of guidelines: bladder pain syndrome. BJU Int. 2018 Nov;122(5):729-743. doi: 10.1111/bju.14399. Epub 2018 Jun 13. PMID 29777618
- [Result] Cox A, Golda N, Nadeau G, Curtis Nickel J, Carr L, Corcos J, Teichman J. CUA guideline: Diagnosis and treatment of interstitial cystitis/bladder pain syndrome. Can Urol Assoc J. 2016 May-Jun;10(5-6):E136-E155. doi: 10.5489/cuaj.3786. Epub 2016 May 12. No abstract available. PMID 27790294